CLINICAL TRIAL: NCT04835662
Title: Engaging Fathers for Improving Dietary Diversity in Kaduna State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20575
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-02

CONDITIONS: Complementary Feeding
Keywords: Minimum dietary diversity; Minimum meal frequency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complementary feeding promotion (Other): Intervention
  Interventions: Behavioral: Complementary feeding promotion

INTERVENTIONS:
Behavioral: Complementary feeding promotion — The intervention engaged fathers through community meetings, religious services, and mobile phone text and voice messages. Mothers received home visits from community health extension workers (CHEWs), which fathers also could attend. Social behavior change communication materials included TV and radio messages, sermon guides, counseling cards, pamphlets, posters, and feeding bowls.

SUMMARY:
The purpose of this study was to evaluate an intervention to engage fathers in supporting the dietary diversity and other complementary feeding practices of their young children.

DETAILED DESCRIPTION:
This was pre-post study designed to measure changes in complementary feeding practices and document the feasibility and acceptability of an intervention to engage fathers in supporting dietary diversity in Kaduna State, Nigeria. This study was conducted as part of the Alive & Thrive Nigeria program, implemented by FHI 360 and partners. RTI led the design and implementation of the study, with Datametrics Associates Ltd. serving as the data collection partner in Nigeria. The study was carried out in 6 wards (2 urban, 4 rural) of Igabi local government area in Kaduna State. We collected survey data cross-sectionally from 495 cohabiting mothers and fathers of children 6-23 months at baseline and endline. Participants were randomly sampled within 99 clusters selected proportional to population size. The purpose of the surveys was to obtain data on children's complementary feeding, changes in fathers' and mothers' knowledge and attitudes related to complementary feeding, and fathers' support for complementary feeding, and to measure participants' exposure to the intervention components. To measure feasibility and acceptability of the intervention, we conducted 24 in-depth interviews at the end of the intervention with community and religious leaders and Community Health Extension Workers who were involved in implementing the intervention. In addition, we conducted separate focus group discussions with mothers and fathers (8 groups each) at the end of the intervention to learn about changes in social norms related to fathers' engagement in complementary feeding and their experiences with participating in the intervention.

ELIGIBILITY:
Inclusion Criteria: For the surveys, men were eligible to participate in the surveys if they were 18 years of age or older, had a child aged 6 to 23 months, and were living in the same household as the child's mother. Women were eligible to participate if they were aged 18 to 49 years or aged 15 to 17 years and married, had a child aged 6 to 23 months, and were living in the same household as the child's father. For the qualitative component, mothers, fathers, community and religious leaders, and community health extension workers who participated in the intervention were eligible.

-

Exclusion Criteria: Refusal to participate or provide consent.

-

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Men were eligible to participate in the surveys if they were 18 years of age or older, had a child aged 6 to 23 months, and were living in the same household as the child's mother. Women were eligible to participate if they were aged 18 to 49 years or aged 15 to 17 years and married, had a child aged 6 to 23 months, and were living in the same household as the child's father
Enrollment: 2168 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Minimum dietary diversity | 24 hours
  The proportion of children 6-23 months who consumed at least 4 food groups on the previous day (World Health Organization indicator definition)

SECONDARY OUTCOMES:
Minimum feeding frequency | 24 hours
  The proportion of children 6-23 months who consumed minimum number of meals by age group and breastfeeding status (WHO indicator definition)
Minimum acceptable diet | 24 hours
  Proportion of children 6-23 months with both minimum dietary diversity and minimum meal frequency (WHO indicator definition)
Consumption of specific food group | 24 hours
  Proportion of children 6-23 months who consumed each of the 7 food groups that make up the dietary diversity indicator

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Flax, Principal Investigator — RTI International
Locations (1):
- Alive and Thrive, Kaduna, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
The data will be open
Time Frame: January 31, 2022

REFERENCES:
- [Derived] Allotey D, Flax VL, Ipadeola AF, Kwasu S, Adair LS, Valle CG, Bose S, Martin SL. Fathers' Complementary Feeding Support Strengthens the Association Between Mothers' Decision-Making Autonomy and Optimal Complementary Feeding in Nigeria. Curr Dev Nutr. 2022 Jun 2;6(7):nzac098. doi: 10.1093/cdn/nzac098. eCollection 2022 Jul. PMID 35854939
- [Derived] Flax VL, Ipadeola A, Schnefke CH, Kwasu S, Mikail AA, Bose S, Brower AO, Edwards S. Complementary Feeding Social and Behavior Change Communication for Fathers and Mothers Improves Children's Consumption of Fish and Eggs and Minimum Meal Frequency in Kaduna State, Nigeria. Curr Dev Nutr. 2022 Apr 8;6(5):nzac075. doi: 10.1093/cdn/nzac075. eCollection 2022 May. PMID 35669047